CLINICAL TRIAL: NCT04920201
Title: The Effect of Exercise With Wearable Walking Assist Robot in Various Environments in Healthy Adults
Brief Title: The Effect of Exercise With Wearable Walking Assist Robot in Various Environments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yun-Hee Kim, Dr., Ph.D., Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-03-052
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Aging
Keywords: wearable hip assist robot

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single masking (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Over-ground walking without GEMS-H (Experimental)
  Interventions: Other: Over-ground walking without GEMS-H
- Over-ground walking with GEMS-H with resist mode (Experimental)
  Interventions: Device: Over-ground walking with GEMS-H with resist mode
- Stair ascent with GEMS-H with assist mode (Experimental)
  Interventions: Device: Stair ascent with GEMS-H with assist mode
- Incline walking with GEMS-H with assist mode (Experimental)
  Interventions: Device: Incline walking with GEMS-H with assist mode

INTERVENTIONS:
Other: Over-ground walking without GEMS-H — Over-ground walking without GEMS-H (30 min per session, at least 3 times per weeks, total 10 sessions)
  Arms: Over-ground walking without GEMS-H
Device: Over-ground walking with GEMS-H with resist mode — Over-ground walking with GEMS-H with resist mode (30 min per session, at least 3 times per weeks, total 10 sessions)
  Arms: Over-ground walking with GEMS-H with resist mode
Device: Stair ascent with GEMS-H with assist mode — Stair ascent with GEMS-H with assist mode (30 min per session, at least 3 times per weeks, total 10 sessions)
  Arms: Stair ascent with GEMS-H with assist mode
Device: Incline walking with GEMS-H with assist mode — Incline walking with GEMS-H with assist mode (30 min per session, at least 3 times per weeks, total 10 sessions)
  Arms: Incline walking with GEMS-H with assist mode

SUMMARY:
This single-blinded, randomized, controlled trial includes 60 healthy adults. The participants were randomized to four different groups. The first group performed over-ground walking without GEMS-H, the second group performed over-ground walking with GEMS-H applied resistance mode, the third group performed stair ascent with GEMS-H applied assist mode, and the fourth group were designated as the group that performed inclined gait with GEMS-H applied assist mode on a treadmill. Each group is divided in 15 participants.

DETAILED DESCRIPTION:
At the first visit, the subjects are fully informed of the study if appropriate after determining whether they meet the selection criteria. If the subjects meet the selection criteria, the participants were randomized to four different groups. The first group performed over-ground walking without GEMS-H, the second group performed over-ground walking with GEMS-H with resistance mode, the third group performed stair ascent with GEMS-H with assist mode, and the fourth group were designated as the group that performed inclined gait with GEMS-H with assist mode on a treadmill. Each group is divided in 15 participants. Each group completed 30 minutes exercise at least three times per week (total 10 sessions). All measurements were conducted before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 50 to less than 85 years without a history of central nervous system disease

Exclusion Criteria:

* Those who have difficulty walking independently due to problems such as visual field defects or fractures
* Those with severe arthritis or orthopedic problems limiting passive range of motion (ROM) of the lower extremities (knee flexion contracture >10°, knee flexion ROM <90°, hip flexion contracture >25°, ankle plantar flexion contracture >15°)
* Those who have difficulty understanding the exercise program due to severe cognitive decline (Korean-Mini-Mental State Examination, K-MMSE≤10)
* Those who have difficulty participating in exercise programs due to adult diseases such as uncontrolled hypertension and diabetes
* Those who are at risk of falling while walking due to severe dizziness
* Those who are less than 140 cm or more than 185 cm in height that is not suitable size for the wearing of the walking assistance robot
* Those who are overweight based on body mass index (BMI) 35 or higher

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline performance on gait speed after the intervention | Baseline, After the intervention(day12)
  Measure of self selected speeds by measuring the time it takes an individual to walk 10 meters. To perform the test, patient walks 10 meters (33 ft) and the time is measured when the leading foot crosses the start line and the finish line. The instructions are: "Please walk this distance at your normal pace when I say go."

SECONDARY OUTCOMES:
Change from baseline performance on muscle strength after the intervention | Baseline, After the intervention(day12)
  All subjects underwent measurements of muscle strength of lower extremity by using Commander Echo Muscle Tester (measures in lb, kg, N)
Change from baseline performance on Short Physical Performance Battery (SPPB) after the intervention | Baseline, After the intervention(day12)
  The Short Physical Performance Battery (SPPB) is a series of tests used to evaluate lower extremity function and mobility.
Change from baseline performance on Functional Reach Test (FRT) after the intervention | Baseline, After the intervention(day12)
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task.
Change from baseline performance on Four Square Step Test (FSST) after the intervention | Baseline, After the intervention(day12)
  Four Square Step Test (FSST) is a test of dynamic balance and coordination that clinically assesses the participant's ability to step over objects forward, sideways, and backwards.
Change from baseline performance on Berg Balance Scale (BBS) after the intervention | Baseline, After the intervention(day12)
  Berg Balance Scale (BBS) is a 14-item objective measure that assesses static balance and fall risk in adults.
Change from baseline performance on Timed Up and Go test (TUG) after the intervention | Baseline, After the intervention(day12)
  The Timed Up and Go test (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Change from baseline performance on Geriatric Depression Scale (GDS) after the intervention | Baseline, After the intervention(day12)
  The Geriatric Depression Scale (GDS) is a self-report measure of depression.
Change from baseline performance on EuroQol 5 Dimensions (EQ-5D) after the intervention | Baseline, After the intervention(day12)
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change from baseline performance on Fall Efficacy Scale-Korea (FES-K) after the intervention | Baseline, After the intervention(day12)
  The Falls Efficacy Scale (FES) is a ten-item test rated on a 10-point scale from not confident at all to completely confident.
Change from baseline performance on metabolic energy expenditure after the intervention | Baseline, After the intervention(day12)
  All subjects underwent measurements respiratory metabolism energy during treadmill walking at a comfortable speed for 5 minutes. It assess the change of metabolic energy expenditure using a portable cardiopulmonary metabolic system (K5, Rome, Italy).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea